CLINICAL TRIAL: NCT04361994
Title: The GErman Italian Spanish Takotsubo (GEIST) Registry
Acronym: GEIST
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. med. Ingo Eitel (Other)
Collaborators: University of Foggia (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Ingo Eitel, Director, University of Luebeck
Organization: University of Luebeck (Other)
Other Study IDs: 00
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Takotsubo Syndrome
MeSH Terms: conditions — Takotsubo Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
GEIST is a multicenter, international observational registry of patients with Takotsubo syndrome. Data regarding the clinical profile (demographic characteristics, clinical presentation, laboratory measures, electrocardiography /echocardiography / coronary angiography parameters, treatment and medication), in-hospital course and complications and short-/long-term outcome are collected prospectively and retrospectively to increase the understanding of the disease.

DETAILED DESCRIPTION:
The open-ended, multicenter, international GEIST registry collects data from patients with Takotsubo syndrome during the index hospitalization and follow-up. Furthermore, long-term outcome data are acquired with structured telephone interviews, in case patients do not undergo regular outpatient visits in the participating study centers. The GEIST registry retrospectively includes data, which have already been collected, and prospectively continues to enroll patients with newly diagnosed Takotsubo syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Takotsubo syndrome

Exclusion Criteria:

* Non

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed according to the current diagnostic recommendations at the time of clinical presentation
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Day 0
  All-cause mortality (in-hospital, short-term, long-term)
All-cause mortality | 3 Month
  All-cause mortality (in-hospital, short-term, long-term)
All-cause mortality | 6 Month
  All-cause mortality (in-hospital, short-term, long-term)

SECONDARY OUTCOMES:
In-Hospital complications | Day 0
  Cardiogenic shock, pulmonary edema, death, life-threatening arrhythmias, ventricular thrombus formation, right ventricular involvement

CONTACTS AND LOCATIONS:
Locations (2):
- Universität zu Lübeck, Lübeck, Schleswig-Holstein, Germany
- University of Foggia, Foggia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raposeiras-Roubin S, Santoro F, Arcari L, Vazirani R, Novo G, Uribarri A, Enrica M, Lopez-Pais J, Guerra F, Alfonso F, Patz T, Fernandez-Cordon C, Montisci R, Corbi-Pascual M, Marchetti MF, Almendro M, Cacciotti L, Vedia O, El-Battrawy I, Blanco-Ponce E, Brunetti ND, Akin I, Martinez-Selles M, Thiele H, Stiermaier T, Eitel I, Nunez-Gil IJ; GEIST Researchers. Beta-Blockers and Long-Term Mortality in Takotsubo Syndrome: Results of the Multicenter GEIST Registry. JACC Heart Fail. 2025 May;13(5):815-825. doi: 10.1016/j.jchf.2024.11.015. Epub 2025 Feb 5. PMID 39918532
- [Derived] Santoro F, Stiermaier T, Nunez Gil IJ, El-Battrawy I, Patz T, Cacciotti L, Guerra F, Novo G, Musumeci B, Volpe M, Mariano E, Caldarola P, Montisci R, Ragnatela I, Cetera R, Vazirani R, Lluch C, Uribarri A, Corbi-Pascual M, Conty Cardona DA, Akin I, Barbato E, Thiele H, Brunetti ND, Eitel I, Arcari L. Renin angiotensin system inhibitors and outcome in patients with takotsubo syndrome: A propensity score analysis of the GEIST registry. Am Heart J. 2024 Dec;278:127-138. doi: 10.1016/j.ahj.2024.08.019. Epub 2024 Sep 10. PMID 39260785
- [Derived] El-Battrawy I, Santoro F, Nunez-Gil IJ, Patz T, Arcari L, Abumayyaleh M, Guerra F, Novo G, Musumeci B, Cacciotti L, Mariano E, Caldarola P, Parisi G, Montisci R, Vitale E, Volpe M, Corbi-Pasqual M, Martinez-Selles M, Almendro-Delia M, Sionis A, Uribarri A, Thiele H, Brunetti ND, Eitel I, Akin I, Stiermaier T. Age-Related Differences in Takotsubo Syndrome: Results From the Multicenter GEIST Registry. J Am Heart Assoc. 2024 Feb 20;13(4):e030623. doi: 10.1161/JAHA.123.030623. Epub 2024 Feb 13. PMID 38348805
- [Derived] Stiermaier T, Walliser A, El-Battrawy I, Patz T, Mezger M, Rawish E, Andres M, Almendro-Delia M, Martinez-Selles M, Uribarri A, Perez-Castellanos A, Guerra F, Novo G, Mariano E, Musumeci MB, Arcari L, Cacciotti L, Montisci R, Akin I, Thiele H, Brunetti ND, Nunez-Gil IJ, Santoro F, Eitel I. Happy Heart Syndrome: Frequency, Characteristics, and Outcome of Takotsubo Syndrome Triggered by Positive Life Events. JACC Heart Fail. 2022 Jul;10(7):459-466. doi: 10.1016/j.jchf.2022.02.015. Epub 2022 May 4. PMID 35772855
- [Derived] El-Battrawy I, Santoro F, Stiermaier T, Moller C, Guastafierro F, Novo G, Novo S, Mariano E, Romeo F, Romeo F, Thiele H, Guerra F, Capucci A, Giannini I, Brunetti ND, Eitel I, Akin I. Incidence and Clinical Impact of Right Ventricular Involvement (Biventricular Ballooning) in Takotsubo Syndrome: Results From the GEIST Registry. Chest. 2021 Oct;160(4):1433-1441. doi: 10.1016/j.chest.2021.04.072. Epub 2021 May 27. PMID 34052189